CLINICAL TRIAL: NCT05473715
Title: A Parallel-group Phase 4, Open-label, Two-arm Study to Assess the Safety and Efficacy of Intravitreal (IVT) Aflibercept With Proactive Customized Treatment Intervals in Patients ≥50 Years of Age With No Fluid Due to Choroidal Neovascularization (CNV) Lesions Secondary to Neovascular (Wet) Age-related Macular Degeneration (nAMD) Following Treatment Initiation With Aflibercept
Brief Title: A Study to Learn How Well Aflibercept Injected Into the Eye Works and How Safe it is When Given in Customized Treatment Intervals in Patients With an Eye Disease Called Neovascular Age-related Macular Degeneration After Start of Treatment
Acronym: XPAND
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to administrative reasons not related to efficacy or safety.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21912; 2022-000690-73 (EudraCT Number)
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Neovascular (Wet) Age-related Macular Degeneration
Keywords: Aflibercept; Anti-vascular endothelial growth factor; Treatment interval extension
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Customized treatment interval (Experimental): After the initial study injection at baseline, participants will receive their next study injection at Week 16. Participants in this study arm will also be issued a home monitoring device, which will allow for regular OCT monitoring (at least 5 times a week) at home.
  Interventions: Drug: Aflibercept(BAY86-5321, Eylea)
- Treat and extend (T&E) 2 week adjustment (Active Comparator): Participants will receive treatment in intervals maintained (8 weeks) or adjusted in 2 weeks increments each time (up to a maximum of 16 weeks and minimum of 4 weeks), as long as all extension/shortening criteria are met.
  Interventions: Drug: Aflibercept(BAY86-5321, Eylea)

INTERVENTIONS:
Drug: Aflibercept(BAY86-5321, Eylea) — 2mg, intravitreal (IVT) injection

SUMMARY:
Researchers are looking for a better way to treat people who have neovascular (wet) age-related macular degeneration (nAMD or wet AMD). In people with wet AMD, the body makes too much of a protein called vascular endothelial growth factor (VEGF). This causes too many blood vessels to grow in the area of sharpest vision in the eye, called macula. Fluid buildup due to leakage from these vessels can damage the macula, leading to vision problems such as blurring or a blind spot in the central (straight ahead) vision needed for reading or face recognition or car driving. Wet AMD is common in people aged 50 and older.

The study treatment intravitreal aflibercept (also called BAY865321) is injected into the eye. It works by blocking the VEGF protein and thus reduces blood vessel growth. It has already been approved for patients with wet AMD to be given as intravitreal injection monthly at start and then every 8 weeks or longer. Repeated injections of aflibercept prevent worsening of vision but place a burden on the patient.

Doctors try to increase the time between injections (treatment interval) in routine clinical practice based on individual patient needs. This is called treat and extend (T&E). Treatment intervals are stepwise extended or shortened depending on how the treatment works. This is checked with optical coherence tomography (OCT), an imaging technique used to observe relevant changes in the eye.

The main purpose of this study is to learn how well aflibercept works if treatment intervals are extended faster (timepoint of extension is the same for both treatments arms), compared to standard T&E regimen in people with wet AMD in a preselected patient population with no fluid after treatment initiation.

To answer this, researchers will assess changes in vision called best corrected visual acuity (BCVA) between study start and after 36 weeks. Changes will then be compared between participants whose treatment intervals were extended early and those on standard T&E regimen.

All participants will receive 2 mg aflibercept as intravitreal injection for up to 52 weeks in intervals of every 4 to 16 weeks.

Each participant will be in the study for up to 56 weeks. During this time 4 visits to the study site are set for all participants. The other visits are set individually. A final phone call is planned 3 days after treatment at the end of study.

During the study, the doctors and their study team will:

* check patients' eye health using various eye examination techniques (slit lamp microscopy, OCT, and ophthalmoscopy) that may necessitate eye drops to widen the pupil)
* measure patients' eye vision (BCVA)
* do physical examinations
* check vital signs
* ask the participants questions about how they are feeling and what adverse events they are having.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

In addition, participants in the fast extension arm will be provided with a home monitoring OCT device.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and able to read (or if unable to read due to visual impairment, be read to verbatim by the person administering the informed consent or a family member), understand, and willing to sign the informed consent form (ICF).
* Men and women ≥50 years of age.
* At treatment initiation, active macular neovascular lesions secondary to nAMD (Patients with polypoidal choroidal vasculopathy or retinal angiomatous proliferation are eligible to participate in the study, and their condition should be captured in the electronic case report form [eCRF]).
* Treatment initiation with 3 × monthly IVT aflibercept injections (Weeks -16, -12, and -8 to planned study baseline visit) resulting in absence of any fluid at week -8.
* ETDRS BCVA of at least 25 letters (20/320 Snellen equivalent) in the study eye at screening visit.
* Willing, committed, and able to return for all clinic visits and complete all study-related procedures.
* Able to use the provided monitoring device and willing to perform 5 × weekly self-assessments in the Investigator's opinion.
* Women and men of reproductive potential must agree to use adequate contraception when sexually active. This applies for the time period between signing of the ICF and 3 months after the last administration of study drug.

Exclusion Criteria:

* Any contraindication to IVT anti-vascular endothelial growth factor (VEGF) treatment or treatment with Eylea® as detailed in the Summary of Product Characteristics (SmPC).
* Any prior ocular (in the study eye) or systemic treatment (including investigational agents) or surgery for nAMD, except the 3 × monthly IVT aflibercept injections required for treatment initiation and dietary supplements or vitamins.
* Any presence of intraretinal and subretinal fluid.
* Any ocular or systemic condition expected to interfere with study outcomes and procedures, including but not limited to:

  * Scar, fibrosis or other lesions (e.g., retinal pigment epithelium [RPE] tears, macular hole stage 2 or above and others) involving the center of the macula in the study eye.
  * Clinically relevant opacities or conditions involving the optic media including cataract, corneal dystrophies or s.p. corneal transplant in the study eye.
  * Uncontrolled glaucoma (defined as IOP ≥25 mm Hg despite treatment with antiglaucoma medication) in the study eye or prior trabeculectomy or other filtration surgery in the study eye.
  * Intraocular surgery, periocular surgery, or cataract surgery within 90 days before Day 1 in the study eye, except the IVT aflibercept injections required for treatment initiation and any history of vitrectomy, retinal radiation therapy, retinal detachment or treatment or surgery for retinal detachment in the study eye.
  * Aphakia or pseudophakia with absence of posterior capsule (unless as a result of an yttrium aluminum garnet posterior capsulotomy) in the study eye.
* Participation as a patient in any clinical study within 12 weeks before screening.
* Close affiliation with the investigational site; e.g., a close relative of the Investigator, dependent person (e.g., employee or student of the investigational site).
* Previously screen failed patients for this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (2):
  - Retina Center of Ottawa, Ottawa, Ontario
  - GOGiunta ophtalmologie, Sherbrooke, Quebec
- Bristol Eye Hospital, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/21912
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrolled participants in 2 countries, between 25 Apr 2023 (first participant first visit) and 11 Jul 2023 (termination date).
Pre-assignment Details: Four participants were screened; 3 were randomized and treated.
Groups:
- Customized Treatment Interval: After the initial study injection at baseline, participants received their next study injection at Week 16. Participants in this study arm were also issued a home monitoring device, which allowed for regular OCT monitoring (at least 5 times a week) at home.
- Standard T&E: Participants received treatment in intervals maintained (8 weeks) or adjusted in 2 weeks increments each time (up to a maximum of 16 weeks and minimum of 4 weeks), as long as all extension/shortening criteria were met.
Period: Overall Study
Arm/Group | Customized Treatment Interval | Standard T&E
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Trial terminate | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Customized Treatment Interval | Standard T&E | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Best-corrected Visual Acuity (BCVA) (Early Treatment Diabetic Retinopathy Study [ETDRS] Letters)
Description: Visual function was assessed using the ETDRS protocol (Early Treatment Diabetic Retinopathy Study Research Group. 1985). Visual acuity examiners must be certified to ensure consistent measurement of BCVA.
Time Frame: Approximately 11 weeks
Population: The study was terminated before any participant reached primary completion (Week 36), therefore no analyses were performed.
Arm/Group | Customized Treatment Interval | Standard T&E
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Intravitreal (IVT) Aflibercept Injections
Description: Participant took aflibercept on study eye.
Time Frame: Approximately 11 weeks
Population: The study was terminated before any participant reached either primary completion (Week 36) or study completion (Week 52), therefore no analyses were performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Customized Treatment Interval | Standard T&E
Number analyzed (Participants) | 2 | 1
Participants
  0 aflibercept injection | 1 | 0
  1 aflibercept injection | 1 | 1

3. Secondary Outcome: Number of Patients Achieving Pre-defined Treatment Intervals
Description: Pre-defined treatment intervals are: ≥4, ≥8, ≥10, ≥12¸ ≥14, and 16 weeks.
Time Frame: Approximately 11 weeks
Population: The study was terminated before any participant reached study completion (Week 52), therefore no analyses were performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Customized Treatment Interval | Standard T&E
Number analyzed (Participants) | 2 | 2
Participants | NA — The study was terminated before any participant took the second injection. | NA — The study was terminated before any participant took the second injection.

4. Secondary Outcome: Change in BCVA (ETDRS Letters)
Description: as for outcome 1
Time Frame: Approximately 11 weeks
Population: as for outcome 3
Arm/Group | Customized Treatment Interval | Standard T&E
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: AEs that occurred or worsened after the first injection of study drug and no later than 30 days after the last injection of study drug was considered as treatment-emergent adverse events (TEAEs).
Time Frame: Approximately 11 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Customized Treatment Interval | Standard T&E
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: After the first injection of study drug and no later than 30 days after the last injection of study drug, up to 78 days. Adverse event reporting for the all-cause mortality considers all deaths that occurred at any time during the study before the last contact, up to 78 days.
Arm/Group | Customized Treatment Interval | Standard T&E
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

LIMITATIONS AND CAVEATS:
The trial was terminated due to administrative reasons not related to efficacy or safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/15/NCT05473715/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT05473715/SAP_001.pdf